CLINICAL TRIAL: NCT00587756
Title: One-Stage Ultrasound-Guided Hepatectomy for Multiple Bilobar Colorectal Metastases: a Feasible and Effective Alternative to Two-Stage Hepatectomy
Brief Title: Alternative to Two-Stage Hepatectomy
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: Fondazione Humanitas per la Ricerca (Other)
Responsible Party: Prof. Guido Torzilli, University of Milan, Istituto Clinico Humanitas - IRCCS
Other Study IDs: MTX-1STAGE; MTX-CRC-1STAGE
Record Dates: First submitted 2008-01-03; First posted 2008-01-07 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: intraoperative ultrasonography; colorectal liver metastases; hepatectomy; portal vein embolization; Liver
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Prospective cohort of consecutive patients who undergo surgery for colorectal cancer liver metastases
  Interventions: Procedure: One-stage ultrasound guided hepatectomy

INTERVENTIONS:
Procedure: One-stage ultrasound guided hepatectomy — Surgical strategy was based on tumor-vessel relationship at intraoperative ultrasonography (IOUS)and on findings at color-Doppler IOUS.

SUMMARY:
Two-stage hepatectomy with or without portal vein embolization allows to treat multiple bilobar metastases expanding surgical indications for these patients. However, it has some related drawbacks: two operations are needed, and some patients do not complete the treatment strategy for disease progression. Using experience gained from our ultrasound guided resection policy we explored the safety and effectiveness of one-stage surgical procedures in patients otherwise recommended for the two-stage approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with resectable colorectal cancer liver metastases (CLM)
2. 4 or more lesions
3. Bilobar involvement of the liver
4. Contact or close adjacency (less than 0.5 cm) of at least one CLM with major intrahepatic vascular structures (1st or 2nd order portal branches and/or hepatic vein at caval confluence).

Exclusion Criteria:

1. Patients with 3 or less resectable CLM
2. Patients with 4 or more resectable CLM but nor bilobar
3. Patients with 4 or more bilobar resectable CLM without any lesion presenting condition of point 4 of the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients carriers of colorectal cancer liver metastases
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2001-09; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the safety of the procedure. To this purpose we studied morbidity, mortality, amount of blood loss, rate of blood transfusions, and postoperative trend of liver function tests. | 30-day and 90-day postoperatively

SECONDARY OUTCOMES:
The secondary outcome measure was the reliability of the procedure from an oncological standpoint. For this purpose we studied the rate of true local recurrence (cut-edge) after a minimum follow-up of 6 months. | Minimum Follow-up of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — University of Milan, Istituto Clinico Humanitas - IRCCS
Locations (1):
- Istituto Clinico Humanitas - Irccs, Rozzano - Milano, Italy

REFERENCES:
- [Background] Adam R, Laurent A, Azoulay D, Castaing D, Bismuth H. Two-stage hepatectomy: A planned strategy to treat irresectable liver tumors. Ann Surg. 2000 Dec;232(6):777-85. doi: 10.1097/00000658-200012000-00006. PMID 11088072
- [Background] Jaeck D, Oussoultzoglou E, Rosso E, Greget M, Weber JC, Bachellier P. A two-stage hepatectomy procedure combined with portal vein embolization to achieve curative resection for initially unresectable multiple and bilobar colorectal liver metastases. Ann Surg. 2004 Dec;240(6):1037-49; discussion 1049-51. doi: 10.1097/01.sla.0000145965.86383.89. PMID 15570209
- [Background] Torzilli G, Montorsi M, Donadon M, Palmisano A, Del Fabbro D, Gambetti A, Olivari N, Makuuchi M. "Radical but conservative" is the main goal for ultrasonography-guided liver resection: prospective validation of this approach. J Am Coll Surg. 2005 Oct;201(4):517-28. doi: 10.1016/j.jamcollsurg.2005.04.026. PMID 16183489
- [Background] Torzilli G, Montorsi M, Del Fabbro D, Palmisano A, Donadon M, Makuuchi M. Ultrasonographically guided surgical approach to liver tumours involving the hepatic veins close to the caval confluence. Br J Surg. 2006 Oct;93(10):1238-46. doi: 10.1002/bjs.5321. PMID 16953487
- [Background] Torzilli G, Del Fabbro D, Palmisano A, Donadon M, Bianchi P, Roncalli M, Balzarini L, Montorsi M. Contrast-enhanced intraoperative ultrasonography during hepatectomies for colorectal cancer liver metastases. J Gastrointest Surg. 2005 Nov;9(8):1148-53; discussion 1153-4. doi: 10.1016/j.gassur.2005.08.016. PMID 16269386